CLINICAL TRIAL: NCT02740335
Title: A Phase III, Randomized, Double-blind, Multicenter Study to Assess the Efficacy and Safety of OCTAPLEX, a Four-factor Prothrombin Complex Concentrate (4F-PCC), Compared to the 4F-PCC Beriplex® P/N (Kcentra), for the Reversal of Vitamin K Antagonist (VKA) Induced Anticoagulation in Patients Needing Urgent Surgery With Significant Bleeding Risk.
Brief Title: Study of Octaplex, a Four-factor Prothrombin Complex Concentrate (4F-PCC) and Beriplex® P/N (Kcentra) for the Reversal of Vitamin K Antagonist (VKA) Induced Anticoagulation in Patients Needing Urgent Surgery With Significant Bleeding Risk.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: LEX-209
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Significant Bleeding Risk
Keywords: anticoagulant reversal; urgent surgery; invasive procedures; vitamin K; prothrombin complex concentrate; four-factor prothrombin complex concentrate (4F-PCC)
MeSH Terms: conditions — Hemophilia B | interventions — prothrombin complex concentrates; Factor IX; factor IX, factor VII, factor X, prothrombin drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Octaplex (Experimental): Participants to receive1 Octaplex infusion intravenously
  Interventions: Drug: Octaplex
- Beriplex P/N (Kcentra) (Active Comparator): Participants to receive1 Kcentra infusions intravenously
  Interventions: Drug: Beriplex P/N (Kcentra)

INTERVENTIONS:
Drug: Octaplex — OCTAPLEX will be administered by intravenous infusion at a rate of 0.12 mL/kg/min (~3 units/kg/min), up to a maximum rate of 8.4 mL/min (~210 units/min).
  Other Names: 4F PCC; 4 Factor PCC; 4 Factor Prothrombin Concentrate Complex
  Arms: Octaplex
Drug: Beriplex P/N (Kcentra) — Beriplex® P/N (Kcentra) will be administered by intravenous infusion at a rate of 0.12 mL/kg/min (~3 units/kg/min), up to a maximum rate of 8.4 mL/min (~210 units/min).
  Other Names: Kcentra
  Arms: Beriplex P/N (Kcentra)

SUMMARY:
To demonstrate that the efficacy of OCTAPLEX as a reversal agent in patients under Vitamin K Antagonist (VKA) therapy with the need for urgent surgery with significant bleeding risk is clinically non-inferior to that Beriplex® P/N (Kcentra).

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate that the efficacy of OCTAPLEX as a reversal agent in patients under Vitami n K Antagonist (VKA)therapy with the need for urgent surgery with significant bleeding risk is clinically non-inferior to that Beriplex® P/N (Kcentra).

The secondary objective of the study is to investigate the safety and tolerability of OCTAPLEX compared to Beriplex® P/N (Kcentra) in patients under Vitamin K Antagonist (VKA) therapy with the need for urgent surgery with significant bleeding risk.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients at least 18 years of age.
2. Patients currently on oral anticoagulation treatment with VKA of coumadin or warfarin type.
3. Patients being admitted to the hospital or currently hospitalized where:

   * an urgent surgery carrying significant bleeding risk (≥50 mL expected blood loss) is required as part of routine clinical care;
   * the use of oral or parenteral vitamin K alone to reverse anticoagulation is deemed too slow or inappropriate for reversal;
4. Patients with an international normalized ratio (INR) of 2.0 or above at the time of decision to reverse the anticoagulation status.
5. Patients who have given written informed consent and who are able and willing to comply with the procedures described in the study protocol.

Exclusion Criteria

1. Patients with a life expectancy of less than 48 hours per physician's judgment (e.g. patients with a Glasgow Coma Scale equal to 3 or a Head Abbreviated Injury Score of 6, patients requiring continuous inotropic or pressor support, and patients whose status is post cardiac arrest).
2. Patients for whom the planned surgery or procedure is commonly associated with a very low bleeding risk (e.g. catheter placement, gastroscopy).
3. Patients with a history of thromboembolic events (TEEs), myocardial infarction, unstable angina pectoris, critical aortic stenosis, cerebrovascular accident, transient ischemic attack, severe peripheral vascular disease, or disseminated intravascular coagulation within 3 months of enrollment.
4. Patients with a known congenital bleeding disorder.
5. Patients with a known antiphospholipid antibody syndrome.
6. Patients with present or past specific factor inhibitor activity.
7. Patients with thrombocytopenia of <80,000/μL or history of heparin-induced thrombocytopenia.
8. Patients who have received heparin of any type or any non-VKA anticoagulant within 24 hours prior to enrollment into the study or with potential need to receive these medications before completion of hemostasis evaluation at the end of surgery.
9. Patients who have received prothrombin complex concentrates (PCCs), fresh frozen plasma or vitamin K within 72 hours prior to enrollment into the study.
10. Patients with a known history of hypersensitivity to plasma-derived products.
11. Patients with acute major bleeding or polytrauma.
12. Pregnant or nursing women.
13. Patients participating in another interventional clinical study currently or during the past 30 days prior to enrollment into this study.
14. Patients previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, Study Director — International Medical Monitor
Locations (72):
- United States (19):
  - Octapharma Research Site, Aurora, Colorado
  - Octapharma Research Site, New Haven, Connecticut
  - Octapharma Research Site, Miami, Florida
  - Octapharma Research Site, Tampa, Florida
  - Octapharma Research Site, Iowa City, Iowa
  - Octapharma Research Site, Boston, Massachusetts
  - Octapharma Research Site, Rochester, New York
  - Octapharma Research Site, Durham, North Carolina
  - Octapharma Research Site, Cleveland, Ohio
  - Octapharma Research Site, Columbus, Ohio
  - Octapharma Research Site, Dayton, Ohio
  - Octapharma Research Site, Fairborn, Ohio
  - Octapharma Research Site, Pittsburgh, Pennsylvania
  - Octapharma Study Site, Pittsburgh, Pennsylvania
  - Octapharma Research Site (0115), Austin, Texas
  - Octapharma Research Site (0127), Austin, Texas
  - Octapharma Research Site, Dallas, Texas
  - Octapharma Research Site, Round Rock, Texas
  - Octapharma Research Site, Puyallup, Washington
- Belarus (2):
  - Octapharma Research Site, Lesnoy
  - Octapharma Research Site, Minsk
- Bulgaria (5):
  - Octapharma Research Site, Plovdiv
  - Octapharma Research Site, Rousse
  - Octapharma Research Site, Sofia
  - Octapharma Study Site, Sofia
  - Octapharma Research Site, Varna
- Georgia (7):
  - Octapharma Research Site, Batumi
  - Octapharma Research Site, Kutaisi
  - Octapharma Research Site - Tbilisi, Tbilisi
  - Octapharma Research Location - Tbilisi, Tbilisi
  - Octapharma Research Site, Tbilisi
  - Octapharma Research Location, Tbilisi
  - Octapharma Research Site, Zugdidi
- Germany (4):
  - Octapharma Research Site, Berlin
  - Octapharma Research Site, Dresden
  - Octapharma Research Site, Frankfurt am Main
  - Octapharma Research Site, Heidelberg
- Octapharma Research Site, Chisinau, Moldova
- Poland (2):
  - Octapharma Research Site, Bochnia
  - Octapharma Research Site, Lodz
- Romania (5):
  - Octapharma Research Site, Bucharest
  - Octapharma Research Site, Cluj-Napoca
  - Octapharma Research Site, Craiova
  - Octapharma Research Site, Oradea
  - Octapharma Research Site, Timișoara
- Russia (10):
  - Octapharma Research Site, Moscow, Russian Federation
  - Octapharma Research Site, Novosibirsk, Russian Federation
  - Octapharma Research Site, Omsk, Russian Federation
  - Octapharma Research Site, Saint Petersburg, Russian Federation
  - Regional Clinical Hospital, Saratov, Russian Federation
  - Octapharma Research Site, Tver', Russian Federation
  - Octapharma Research Site, Yekaterinburg, Russian Federation
  - Octapharma Research Site, Moscow
  - Octapharma Research Site, Saint Petersburg
  - Octapharma Research Site, Smolensk
- Spain (3):
  - Octapharma Research Site, Barcelona
  - Octapharma Research Site, Palma de Mallorca
  - Octapharma Research Site, Valencia
- Ukraine (14):
  - Octapharma Research Site, Cherkasy
  - Octapharma Research Site, Chernivtsi
  - Octapharma Research Location, Dnipro
  - Octapharma Research Site, Dnipro
  - Octapharma Research Site, Ivano-Frankivsk
  - Octapharma Research Site, Kharkiv
  - Octapharma Research Site, Kropyvnytskyi
  - Octapharma Research Site, Kyiv
  - Octapharma Research Site, Lutsk
  - Octapharma Research Site, Lviv
  - Octapharma Research Site, Odesa
  - Octapharma Research Site, Vinnytsia
  - Octapharma Research Site, Zaporizhzhya
  - Octapharma Research Site, Zhytomyr

REFERENCES:
- [Background] American Society of Anesthesiologists Task Force on Perioperative Blood Transfusion and Adjuvant Therapies. Practice guidelines for perioperative blood transfusion and adjuvant therapies: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Blood Transfusion and Adjuvant Therapies. Anesthesiology. 2006 Jul;105(1):198-208. doi: 10.1097/00000542-200607000-00030. No abstract available. PMID 16810012
- [Background] Campbell P, Roberts G, Eaton V. Managing warfarin therapy in the community. Aust Prescriber 2001; 24:86-89.
- [Background] Cushman M, et al. Clinical Practice Guide on Antithrombotic Drug Dosing and Management of Antithrombotic Drug-Associated Bleeding Complications in Adults, American Society of Hematology, 2014.
- [Background] Gohlke-Barwolf C. [Anticoagulation in surgery, after hemorrhagic complications and in pregnancy]. Z Kardiol. 1998;87 Suppl 4:56-62. German. PMID 9857468
- [Background] Goldstein JN, Refaai MA, Milling TJ Jr, Lewis B, Goldberg-Alberts R, Hug BA, Sarode R. Four-factor prothrombin complex concentrate versus plasma for rapid vitamin K antagonist reversal in patients needing urgent surgical or invasive interventions: a phase 3b, open-label, non-inferiority, randomised trial. Lancet. 2015 May 23;385(9982):2077-87. doi: 10.1016/S0140-6736(14)61685-8. Epub 2015 Feb 27. PMID 25728933
- [Background] Hwang IK, Shih WJ, De Cani JS. Group sequential designs using a family of type I error probability spending functions. Stat Med. 1990 Dec;9(12):1439-45. doi: 10.1002/sim.4780091207. PMID 2281231
- [Background] Keeling D, Baglin T, Tait C, Watson H, Perry D, Baglin C, Kitchen S, Makris M; British Committee for Standards in Haematology. Guidelines on oral anticoagulation with warfarin - fourth edition. Br J Haematol. 2011 Aug;154(3):311-24. doi: 10.1111/j.1365-2141.2011.08753.x. Epub 2011 Jun 14. No abstract available. PMID 21671894
- [Background] Lankiewicz MW, Hays J, Friedman KD, Tinkoff G, Blatt PM. Urgent reversal of warfarin with prothrombin complex concentrate. J Thromb Haemost. 2006 May;4(5):967-70. doi: 10.1111/j.1538-7836.2006.01815.x. PMID 16689743
- [Background] Makris M, Greaves M, Phillips WS, Kitchen S, Rosendaal FR, Preston EF. Emergency oral anticoagulant reversal: the relative efficacy of infusions of fresh frozen plasma and clotting factor concentrate on correction of the coagulopathy. Thromb Haemost. 1997 Mar;77(3):477-80. PMID 9065997
- [Background] Oden A, Fahlen M. Oral anticoagulation and risk of death: a medical record linkage study. BMJ. 2002 Nov 9;325(7372):1073-5. doi: 10.1136/bmj.325.7372.1073. PMID 12424167
- [Background] Palareti G, Leali N, Coccheri S, Poggi M, Manotti C, D'Angelo A, Pengo V, Erba N, Moia M, Ciavarella N, Devoto G, Berrettini M, Musolesi S. Bleeding complications of oral anticoagulant treatment: an inception-cohort, prospective collaborative study (ISCOAT). Italian Study on Complications of Oral Anticoagulant Therapy. Lancet. 1996 Aug 17;348(9025):423-8. doi: 10.1016/s0140-6736(96)01109-9. PMID 8709780
- [Background] A randomized trial of anticoagulants versus aspirin after cerebral ischemia of presumed arterial origin. The Stroke Prevention in Reversible Ischemia Trial (SPIRIT) Study Group. Ann Neurol. 1997 Dec;42(6):857-65. doi: 10.1002/ana.410420606. PMID 9403477
- [Background] van Aart L, Eijkhout HW, Kamphuis JS, Dam M, Schattenkerk ME, Schouten TJ, Ploeger B, Strengers PF. Individualized dosing regimen for prothrombin complex concentrate more effective than standard treatment in the reversal of oral anticoagulant therapy: an open, prospective randomized controlled trial. Thromb Res. 2006;118(3):313-20. doi: 10.1016/j.thromres.2005.08.005. Epub 2005 Sep 21. PMID 16182346
- [Background] Yasaka M, Sakata T, Minematsu K, Naritomi H. Correction of INR by prothrombin complex concentrate and vitamin K in patients with warfarin related hemorrhagic complication. Thromb Res. 2002 Oct 1;108(1):25-30. doi: 10.1016/s0049-3848(02)00402-4. PMID 12586128
- [Derived] Sarode R, Goldstein JN, Simonian G, Hinterberger D, Matveev D, Gareis M, Milling TJ Jr. Vitamin K Antagonist Reversal for Urgent Surgery Using 4-Factor Prothrombin Complex Concentrates: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2424758. doi: 10.1001/jamanetworkopen.2024.24758. PMID 39088218

RESULTS

PARTICIPANT FLOW:
Groups:
- Beriplex P/N (Kcentra): Participants to receive1 Kcentra infusion intravenously
  Beriplex P/N (Kcentra): Beriplex® P/N (Kcentra) will be administered by intravenous infusion at a rate of 0.12 mL/kg/min (~3 units/kg/min), up to a maximum rate of 8.4 mL/min (~210 units/min).
Period: Overall Study
Arm/Group | Octaplex | Beriplex P/N (Kcentra)
Started | 105 | 103
Completed | 105 | 103
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Beriplex P/N (Kcentra): Participants to receive 1 Kcentra infusion intravenously
  Beriplex P/N (Kcentra): Beriplex® P/N (Kcentra) will be administered by intravenous infusion at a rate of 0.12 mL/kg/min (~3 units/kg/min), up to a maximum rate of 8.4 mL/min (~210 units/min).
- Total: Total of all reporting groups
Arm/Group | Octaplex | Beriplex P/N (Kcentra) | Total
Number analyzed (Participants) | 105 | 103 | 208
Age, Continuous [Mean (Full Range); unit: Years] | 65.6 [31 to 90] | 66.8 [32 to 92] | 66.2 [31 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 43 | 90
  Male | 58 | 60 | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 105 | 102 | 207
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Pre-Infusion Anticoagulation Therapy [Number; unit: participants]
  Sol. Fraxiparine (nadroparin calcium) | 1 | 0 | 1
  Vitamin K Antagonist | 105 | 103 | 208
History of TEE [Number; unit: participants]
  Presence of Embolic or Thrombotic Event | 13 | 18 | 31
  Absence of Embolic or Thrombotic Event | 92 | 85 | 177
Type of Surgey [Number; unit: participants]
  Cardiothoracic Surgery | 5 | 4 | 9
  Orthopaedic Surgery | 7 | 5 | 12
  Other Surgery Type | 93 | 94 | 187
Estimated Average Blood Loss [Number; unit: participants] — Expected average blood loss in mL during surgery for non-anticoagulated patients undergoing the same type of surgical procedure
  participants
    ≥200 mL | 55 | 50 | 105
    ≥100 mL but <200 mL | 26 | 25 | 51
    ≥50mL but <100 mL | 24 | 28 | 52

OUTCOME MEASURES:

1. Primary Outcome: Hemostatic Efficacy Rating by IEAB
Description: Hemostatic Efficacy rated by the Independent Endpoint Adjudication Committee based on a 1 to 4 point hemostatic efficacy scale, taking into account blood loss and transfusion requirements in the context of the surgery. Hemostatic efficacy was assessed based on objective criteria in the categories 'excellent', 'good', 'moderate', or 'none'. Ratings of 'excellent' and 'good' were considered as 'effective' hemostasis, while ratings of 'moderate' and 'none' were considered as 'ineffective' hemostasis.
Time Frame: At the end of the surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex | Beriplex P/N (Kcentra)
Number analyzed (Participants) | 105 | 103
Participants
  Excellent - 4 | 41 | 50
  Good - 3 | 58 | 47
  Moderate - 2 | 6 | 6
  None - 1 | 0 | 0
  Effective | 99 | 97
  Ineffective | 6 | 6

2. Primary Outcome: Dichotomous Hemostasis Success
Description: To demostrate clinical non-inferiority of treatment with Octaplex to treatment with Beriplex P/N (Kcentra) with respect to hemostatic success. Effective hemostatis includes Excellent and Good ratings, while Ineffective hemostasis includes Moderate, None and missing ratings from Global hemostatic efficacy observed by IEAB
Time Frame: At the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex | Beriplex P/N (Kcentra)
Number analyzed (Participants) | 105 | 103
Participants
  Effective | 99 | 97
  Ineffective | 6 | 6

3. Secondary Outcome: Measuring of International Normalized Ratio (INR) to ≤ 1.5
Description: Number of patients with an international normalized ratio (INR) value of less or equal to 1.5 at 30 min (± 15 min) after the end of infusion.
Time Frame: 30 minutes after the end of infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex | Beriplex P/N (Kcentra)
Number analyzed (Participants) | 105 | 103
Participants
  <=1.5 | 82 | 74
  > 1.5 | 23 | 29
  Missing | 0 | 0

4. Secondary Outcome: Coagulation Factor II Levels
Description: Change in coagulation factor levels from baseline to after the end of infusion using the Hodges-Lehmann Estimator for median differences: o Factor II
  The Hodges-Lehmann Estimator is a method of robust estimation. This estimator is used to give an estimate of the difference between the values in two sets of data. If the two sets of data contain m and n data points respectively, m × n pairs of points (one from each set) can be formed and each pair gives a difference of values. The Hodges-Lehmann estimator for the difference is defined as the median of the m × n differences.
Time Frame: 30 minutes after the end of infusion
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Octaplex | Beriplex P/N (Kcentra)
Number analyzed (Participants) | 105 | 103
mg/dL | 49.5 [37.0 to 76.5] | 51.0 [37.5 to 69.0]

5. Secondary Outcome: Coagulation Factor VII Levels
Description: Change in coagulation factor levels from baseline to after the end of infusion using the Hodges-Lehmann Estimator for median differences: o Factor VII
  The Hodges-Lehmann Estimator is a method of robust estimation. This estimator is used to give an estimate of the difference between the values in two sets of data. If the two sets of data contain m and n data points respectively, m × n pairs of points (one from each set) can be formed and each pair gives a difference of values. The Hodges-Lehmann estimator for the difference is defined as the median of the m × n differences.
Time Frame: 30 minutes after the end of infusion
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Octaplex | Beriplex P/N (Kcentra)
Number analyzed (Participants) | 105 | 103
mg/dL | 35.0 [21.0 to 55.0] | 23.0 [15.0 to 43.0]

6. Secondary Outcome: Coagulation Factor IX Levels
Description: Change in coagulation factor levels from baseline to after the end of infusion using the Hodges-Lehmann Estimator for median differences: o Factor II Factor IX
  The Hodges-Lehmann Estimator is a method of robust estimation. This estimator is used to give an estimate of the difference between the values in two sets of data. If the two sets of data contain m and n data points respectively, m × n pairs of points (one from each set) can be formed and each pair gives a difference of values. The Hodges-Lehmann estimator for the difference is defined as the median of the m × n differences.
Time Frame: 30 minutes after the end of infusion
Measure: Mean (95% Confidence Interval); unit: m/dL
Arm/Group | Octaplex | Beriplex P/N (Kcentra)
Number analyzed (Participants) | 105 | 103
m/dL | 33.0 [17.0 to 56.0] | 31.5 [19.0 to 51.0]

7. Secondary Outcome: Coagulation Factor X Levels
Description: Change in coagulation factor levels from baseline to after the end of infusion using the Hodges-Lehmann Estimator for median differences: o Factor X
  The Hodges-Lehmann Estimator is a method of robust estimation. This estimator is used to give an estimate of the difference between the values in two sets of data. If the two sets of data contain m and n data points respectively, m × n pairs of points (one from each set) can be formed and each pair gives a difference of values. The Hodges-Lehmann estimator for the difference is defined as the median of the m × n differences.
Time Frame: 30 minutes after the end of infusion
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Octaplex | Beriplex P/N (Kcentra)
Number analyzed (Participants) | 105 | 103
mg/dL | 50.0 [35.0 to 73.0] | 63.0 [49.0 to 88.0]

8. Secondary Outcome: Number of Patients Requiring Red Blood Cells (RBC)
Description: Number of patients receiving red blood cells (RBC) during the surgery
Time Frame: At the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Octaplex | Beriplex P/N (Kcentra)
Number analyzed (Participants) | 105 | 103
Participants
  Received RBC | 4 | 3
  Did Not Receive RBC | 101 | 100

ADVERSE EVENTS:
Time Frame: 45 days after surgery
Groups:
- Octaplex: Participants to receive 1 Octaplex infusion intravenously
  Octaplex: OCTAPLEX will be administered by intravenous infusion at a rate of 0.12 mL/kg/min (~3 units/kg/min), up to a maximum rate of 8.4 mL/min (~210 units/min).
Arm/Group | Octaplex | Beriplex P/N (Kcentra)
All-Cause Mortality (participants affected / at risk) | 5/105 | 1/103
Serious Adverse Events (participants affected / at risk) | 13/105 | 6/103
Other Adverse Events (participants affected / at risk) | 86/105 | 80/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octaplex (N=105) | Beriplex P/N (Kcentra) (N=103)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Chronic (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric Haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic Haemmorhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Failure to Anastomose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft Tissue Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ovarian Cancer Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octaplex (N=105) | Beriplex P/N (Kcentra) (N=103)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 5 (5)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Cardiac AEs (Cardiac disorders) | 5 (5) | 7 (7)
Asthenia (General disorders) | 13 (13) | 18 (18)
Catheter Site Related Reaction (General disorders) | 4 (4) | 2 (2)
Hyperthermia (General disorders) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Procedural Pain (Injury, poisoning and procedural complications) | 50 (50) | 50 (50)
Postoperative Wound Complications (Injury, poisoning and procedural complications) | 15 (15) | 15 (15)
Procedural Vomiting (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Suture Related Complication (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Blood Pressure Increase (Investigations) | 0 (0) | 5 (5)
Body Temperature Increase (Investigations) | 0 (0) | 4 (4)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (4) | 7 (7)
Nervous System Disorders (Nervous system disorders) | 6 (6) | 1 (1)
Dysuria (Renal and urinary disorders) | 5 (5) | 2 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Vascular Disorders (Vascular disorders) | 1 (1) | 6 (6)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT02740335/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT02740335/SAP_001.pdf